CLINICAL TRIAL: NCT06447883
Title: Influence of Lifestyle Modification Program on Meaningful Participation and Quality of Life of Independent Taiwanese Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hui-Jen Shyu (Other)
Collaborators: Kaohsiung Medical University (Other)
Responsible Party: Sponsor-Investigator, Hui-Jen Shyu, Principal Investigator, National Taiwan University
Organization: National Taiwan University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KMUHIRB-E(I)-20170158
Record Dates: First submitted 2024-02-15; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Quality of Life

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle modification program (Experimental): The LMP included 12 treatment modules which was administered by the occupational therapist with a national occupational therapist license and a certification from the USC Lifestyle Redesign® course in 2001. The experimental group engaged in 24 weekly group sessions, each lasting approximately 2 hours. Each session started with stretching, followed by knowledge sharing, group discussion, and activities participation which aligned with the session's themes and discussion topics. The four strategies, including didactic presentation, peer exchange, direct experience, and personal exploration, were employed to deliver the treatment module content. Following these strategies, the primary researcher emphasized the connection between participants' personal meanings, individual contexts, and occupations. Afterward, participants were encouraged to formulate a personalized action plan and integrate what they had learnt into their daily routine.
  Interventions: Behavioral: Lifestyle modification program
- Control group (No Intervention): The control group participants were selected from the same community as the experimental group but did not receive the LMP.

INTERVENTIONS:
Behavioral: Lifestyle modification program — The LMP included 12 treatment modules which was administered by the occupational therapist with a national occupational therapist license and a certification from the USC Lifestyle Redesign® course in 2001. The experimental group engaged in 24 weekly group sessions, each lasting approximately 2 hours. Each session started with stretching, followed by knowledge sharing, group discussion, and activities participation which aligned with the session's themes and discussion topics. The four strategies, including didactic presentation, peer exchange, direct experience, and personal exploration, were employed to deliver the treatment module content. Following these strategies, the primary researcher emphasized the connection between participants' personal meanings, individual contexts, and occupations. Afterward, participants were encouraged to formulate a personalized action plan and integrate what they had learnt into their daily routine.
  Arms: Lifestyle modification program

SUMMARY:
The goal of this clinical trial is to compare the differences between health-related quality of life and meaningful participation among two groups.

The main question it aimed to answer are: whether the older adults from experimental group who received 24-week lifestyle modification program would have higher level of health-related quality of life and meaningful participation compared to those who did not receive the program from the control group. Participants in experimental group had to attend in a 24-week lifestyle modification program. Researchers will compare the experimental and control group to see if there were differences between their health-related quality of life and meaningful participation.

DETAILED DESCRIPTION:
This study investigates the impact of a Lifestyle Modification Program (LMP) on the quality of life and meaningful participation of independent Taiwanese older adults. As the global and Taiwanese populations age rapidly, there's an urgent need to address the challenges posed by aging, including deteriorations in physical and mental health that affect independent living and well-being. Inspired by USC's Lifestyle Redesign® Program, this research aimed to adapt and evaluate a similar intervention in a Taiwanese context, considering cultural differences and specific needs.

Participants in the experimental and control groups were required to be over 55 years old, independently living in the community, proficient in Mandarin Chinese or Taiwanese, and showing no overt signs of psychosis or dementia. The study was conducted with ethical approval from Kaohsiung Medical University's IRB, ensuring confidentiality and informed consent.

The experimental group received the LMP which included 12 treatment modules delivered in 24 weekly group sessions, emphasizing active engagement, knowledge sharing, and personal exploration. The intervention aimed to foster psychophysical health, increase daily activity participation, and enhance overall quality of life through a large group format over a shorter timeframe than traditional interventions. The control group participants were selected from the same community without engaged in the LMP.

The study used the SF-36 Taiwan version to measure health-related quality of life and the Taiwanese Meaningful Activity Participation Assessment (T-MAPA) to evaluate the frequency and degree of meaningful participation, and then to compared the changed scores between the two groups in order to examine the efficacy of the LMP. Additionally, individual semi-structured interviews were conducted to acquire qualitative insights into participants' subjective experiences before, during, and after the intervention among the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* over 55 years old
* independently community-dwelling
* proficient in Mandarin Chinese or Taiwanese

Exclusion Criteria:

-show overt signs of psychosis or dementia

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
SF-36 Taiwan version | pre-intervention and immediately after the intervention
  Health-related quality of life (QoL) was measured by the SF-36 Taiwan version, a, standardized, self-report questionnaire commonly used to determine the effect of medical and community-based health intervention. Comprising 36 questions, it gauges self-perceived physical health and mental well-being over the past four weeks across eight domains: Physical Functioning, Role Limitations due to Physical Health Problems (Role-Physical), Bodily Pain, General Health, Vitality, Social Functioning, Role Limitations due to Emotional Problems (Role-Emotional), and Mental Health. Responses within each domain were summed and transformed, generating dimension scores ranging from 0 (poor health) to 100 (good health). The experimental and control groups completed the measurement pre-intervention and immediately after the experimental group received the intervention.
Taiwanese version of the Meaningful Activity Participation Assessment | pre-intervention and immediately after the intervention
  This study assessed the frequency and degree of meaningful participation using the Taiwanese version of the Meaningful Activity Participation Assessment (T-MAPA). This 25-item tool, yields scores ranging from 0 to 300, with higher scores denoting increased meaningful participation over the past three months. Culturally adapted to Taiwan, the T-MAPA has demonstrated robust reliability and validity.The experimental and control groups completed the measurement pre-intervention and immediately after the experimental group received the intervention.
Individual semi-structured interviews | pre-intervention, during the intervention, and immediately after the intervention
  Individual semi-structured interviews were conducted with participants in the experimental group at three stages during the study, including pre-intervention, during the intervention, and immediately after the intervention, each lasting 30 to 90 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No